CLINICAL TRIAL: NCT01486628
Title: A Phase I, Single Dose, Single-centre, Randomized, Double-blind, Placebo-controlled Dose Escalation Study Evaluating Safety, Tolerability and Levodopa Plasma Concentration Following Administration of Subcutaneous Continuously-delivered Levodopa/Carbidopa Solution (ND0612) in Healthy Volunteers
Brief Title: Study of Subcutaneous Continuous Administration of Levodopa/Carbidopa Solution (ND0612) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroDerm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ND0612/001 and 001b
Record Dates: First submitted 2011-12-04; First posted 2011-12-06 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- levodopa and carbidopa (Placebo Comparator)
  Interventions: Drug: ND0612
- Placebo (Placebo Comparator): Saline solution for subcutaneous administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ND0612 — levodopa and carbidopa solution for subcutaneous administration
  Arms: levodopa and carbidopa
Drug: Placebo — Saline solution for SC continuous administration
  Arms: Placebo

SUMMARY:
It will be a single dose, single-center, randomized, double-blind, placebo-controlled dose escalation study of SC continuously-delivered LD/CD solution (ND-0612) for 24 hours in healthy volunteers.

Objectives are to determine:

1. the maximal tolerated dose of SC ND-0612
2. the steady state plasma concentration of LD and CD following SC ND-0612 administration.

Each treatment group will include 6 healthy volunteers. Dosing will be done in a sequential manner.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian males between 18 and 40 years (inclusive) of age
* Normal BMI (18.5-24.9)
* Subjects with negative urinary drugs of abuse, HIV, Hepatitis B or Hepatitis C serology tests
* Subjects must be able to adhere to the protocol requirements
* Subjects must provide written informed consent to participate in the study.

Exclusion Criteria:

* History of significant psychiatric disorder, neurological diseases or sleep disorders
* History of significant systemic diseases, by medical history or tests performed during screening examinations
* Clinically significant laboratory tests at screening
* History of drug or alcohol abuse.
* Allergy to levodopa, carbidopa or any inactive component of the test formulation.
* Subjects with dark skin
* Subjects with skin diseases or neoplasms
* Subjects with narrow-angle glaucoma
* Subjects with significant allergic response to other drugs.
* Presence of clinically significant scars or other skin disorders in the area of placement of the pump.
* Use of any prescription or over-the-counter (OTC) medications
* Subjects who donated blood or received blood, in the last 3 months
* Participation in another clinical trial in the last 30 days
* Subjects which do not have the ability to communicate well or will not adhere to the protocol procedures

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2012-11-22 (Actual); Study Completion 2013-06-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 2 weeks
  The safety and tolerability of ND0612 will be well monitored and will assess the ND0612 effect at various doses in comparison to placebo in the following parameters:
  * Incidence and frequency of local adverse events related to the ND0612 Sc administration.
  * Local safety scoring. In addition, systemic adverse events and withdrawal rates and discontinuations due to adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel